CLINICAL TRIAL: NCT02514018
Title: A Pilot Study to Characterize the Immune Response Induced by a Commercial Varicella Zoster Virus Vaccine in Healthy Adult Females in Nairobi, Kenya.
Brief Title: Pilot Study to Describe Immune Responses of Healthy Women Following Immunization With Varicella Zoster Virus Vaccine
Acronym: KAVI-VZV-001
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Kenyan AIDS Vaccine Initiative - Institute of Clinical Research (KAVI-ICR) (Unknown); University of Nairobi (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr Walter Jaoko, Professor, University of Nairobi
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KAVI-VZV-001
Record Dates: First submitted 2015-06-29; First posted 2015-08-03 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Varicella-Zoster Virus; Immune Activation; HIV Vaccine; Mucosal Immunity
MeSH Terms: conditions — Chickenpox | interventions — Herpes Zoster Vaccine; Chickenpox Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Group (Other): Live-attenuated varicella-zoster virus vaccine (≥ 19,400 Plaque-forming unit - PFU) administered as a single-dose at day 0
  Interventions: Biological: Live-attenuated varicella-zoster virus vaccine
- Delayed Group (Other): Live-attenuated varicella-zoster virus vaccine (≥ 19,400 PFU) administered as a single-dose at day 84 (+/- 3 days)
  Interventions: Biological: Live-attenuated varicella-zoster virus vaccine

INTERVENTIONS:
Biological: Live-attenuated varicella-zoster virus vaccine — Commercial vaccine used to prevent shingles
  Other Names: shingles vaccine; chickenpox vaccine; zoster vaccine; Zostavax® (Merck)

SUMMARY:
The re-activating nature of Varicella Zoster Virus (VZV) may allow life long boosting when used as a vaccine vector in conjunction with HIV to generate durable immunity systemically and at the mucosa. This study aims to characterize mucosal immunity before and after vaccination with a commercial live-attenuated varicella-zoster virus vaccine with respect to immune activation state, mucosal homing properties and VZV-specific effector immune responses in healthy women at low risk for HIV acquisition.

DETAILED DESCRIPTION:
An ideal HIV vaccine should be able to induce an effector specific immune response at the mucosal site which serves as the portal of HIV entry. The use of a persistent replicating viral vector such as Varicella-Zoster Virus (VZV) has great potential to assemble this specific response. Live-attenuated varicella-zoster virus has been used as a vaccine worldwide for over 25 years and has a well-described safety profile. However, its immunogenicity data in the African population are lacking.

The general objective of this study will be to measure the magnitude and kinetics of the effector immune response and immune activation induced by live-attenuated varicella-zoster virus vaccine in a population of Kenyan women. Specifically, the study will measure immune activation in both cervical and rectal mucosae in the context of VZV-effector responses after vaccination and compare the observed immune activation in mucosal tissues and in blood.

A total of 44 healthy women in Nairobi, aged 18-50 years will be recruited into the study, after obtaining their written informed consent. Eligibility to participate in the study will depend on results of laboratory tests, review of medical history, physical examination and answers to questions about HIV risk behaviours.

The study will assess immune responses to both immediate and delayed administration of live-attenuated virus varicella-zoster vaccine in VZV-seropositive individuals. Participants will be randomly divided into 2 groups. Group 1 will receive a single dose of the vaccine at day 0 and Group 2 at day 84. The participants will be followed for a period of 9-12 months after receiving the vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy females, as assessed by a medical history, physical examination and laboratory tests;
2. Aged at least 18 years on the day of screening and no greater than 50 years on the day of the first vaccination.
3. VZV-seropositive, as assessed by the Vitek Immunodiagnostic Assay System (VIDAS) assay.
4. Ability to comply with the study requirements and available for follow-up for the planned duration of the study.
5. In the opinion of the Principal Investigator or designee, the volunteer has understood the information provided and signed the consent document.
6. Willing to undergo HIV testing, HIV counseling and to receive HIV test results three times during the study.
7. For women with potential to become pregnant, willing to use effective contraception or barrier methods, such as oral, patch, injectable, implant, ring contraceptives or intrauterine device to avoid pregnancy during the study (spermicide are not allowed).

Exclusion Criteria:

Any relevant abnormality on history or examination that, in the opinion of the Principal Investigator or designee, is clinically significant, and/or:

1. A high risk for HIV-acquisition defined by the experience of any of the follow situations:

   1. Had unprotected vaginal or anal sex with a known HIV-1-infected person, a person known to be at high risk for HIV or a casual partner (i.e., no continuing, established relationship) within the previous 6 months;
   2. Engaged in sex work for money or drugs within the previous 6 months;
   3. Used injection drugs in the last 12 months;
   4. Abuse of illicit or prescribed drugs, including alcohol;
   5. Acquired one of the following sexually transmitted infection: chlamydia, gonorrhoea and syphilis in the last 12 months;
   6. More than 1 sexual partner within the last 6 months;
   7. New sexual partner within the last 3 months.
2. Persistent or recurrent bacterial vaginosis or vaginal candidiasis unresponsive to therapy (2 consecutive attempts by study team).
3. Confirmed HIV-1 or HIV-2 infection.
4. Any clinically significant acute or chronic medical condition that is considered progressive or, in the opinion of the Principal Investigator or designee, would make the volunteer unsuitable for the study (active or underlying diabetes, gastrointestinal, cardiovascular, malignancy, neurological, psychiatric, metabolic, renal, hepatic, respiratory, auto-immune diseases, psoriasis, primary and acquired immunodeficiency status and rectal problems).
5. Significant laboratory abnormalities, including coagulation (International Normalised Ratio- INR <1.0 or > 1.5).
6. A positive pregnancy test or breast-feeding at screening; for the participants with reproductive potential, unwilling to use an effective method of preventing pregnancy during the study.
7. Receipt of vaccine within the previous 2 months or planned receipt at any time until 6 months after vaccination with live-attenuated VZV vaccine.
8. Receipt of blood transfusion or blood products within the previous 6 months.
9. Participation in another interventional clinical trial currently or within the previous 3 months.
10. History of severe or very severe local or systemic reactogenicity events after vaccination, history of severe or very severe allergic reactions, or history of anaphylactic/anaphylactoid reaction to neomycin.
11. History of toxic shock syndrome.
12. Confirmed diagnosis of acute or chronic hepatitis B virus infection (spontaneous clearance leading to natural immunity, indicated by antibodies to core + antigens, is not an exclusion criterion); confirmed diagnosis of hepatitis C virus infection.
13. Immunosuppressive medications 30 days before or during the study period.
14. Major psychiatric illness including any history of schizophrenia or severe psychosis, bipolar disorder, suicidal attempt or ideation in the previous 3 years.
15. Contra-indication for undergoing a biopsy due to bleeding diathesis, haemorrhoids, mucosal infection at the biopsy site, medication that interfere with clotting (e.g. warfarin or heparin) - both clinical and laboratory.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in the median frequency of cervical CD38+HLA-DR+CD4+T cells after VZV-vaccination as a measure of immune activation | 3 months after VZV-vaccination
  Comparison of the change in the median (Interquartile range - IQR) frequency of cervical CD38+HLA-DR+CD4+T cells between 1) Baseline and 3 months after (for the delayed group), and 2) Before and after 3 months of VZV vaccination (immediate and delayed groups).

SECONDARY OUTCOMES:
Composite measures of immune activation observed in mucosal tissues | 3 months after VZV-vaccination
  Comparison of the change in the median (IQR) expression of activation markers such as CD38, CD69, Ki67 and HLA-DR in mucosal T cells (CD4+ and CD8+ T cells) between 1) Baseline and 3 months after (for the delayed group), and 2) Before and after 3 months of VZV vaccination (immediate and delayed groups)
Composite measures of mucosal homing marker and HIV co-receptors observed in mucosal tissues | 3 months after VZV-vaccination
  Comparison of the change in the median (IQR) expression of α4β7 and CCR5 in mucosal CD4+T cells between 1) Baseline and 3 months after (for the delayed group), and 2) Before and after 3 months of VZV vaccination (immediate and delayed groups)
Mucosal level of inflammation (including IL-1β, IL-6 and IL8) | 3 months after VZV-vaccination
Composite measures of immune activation observed in blood | 3 months after VZV-vaccination
  Comparison of the change in the median (IQR) expression activation markers such as CD38, CD69, Ki67 and HLA-DR in systemic T cells (CD4+ and CD8+ T cells) between 1) Baseline and 3 months after (for the delayed group), and 2) Before and after 3 months of VZV vaccination (immediate and delayed groups)
Composite measures of mucosal homing marker and HIV co-receptors observed in blood | 3 months after VZV-vaccination
  Comparison of the change in the median (IQR) expression of α4β7 and CCR5 in systemic CD4+T cells between 1) Baseline and 3 months after (for the delayed group), and 2) Before and after 3 months of VZV vaccination (immediate and delayed groups).
Plasma level of inflammation (including IL-1β, IL-6 and IL8) | 3 months after VZV-vaccination
Frequency and function of mucosal VZV-specific immune cells (including CD8+ and CD4+ T cell subsets) | Longidudinally througout the study (up to 12 months)
Concentration of mucosal VZV-specific antibodies (IgG and IgA) | Longidudinally througout the study (up to 12 months)
Frequency and function of systemic VZV-specific immune cells (including CD8+ and CD4+ T cell subsets) | Longidudinally througout the study (up to 12 months)
Concentration of systemic VZV-specific antibodies (IgG and IgA) | Longidudinally througout the study (up to 12 months)

OTHER OUTCOMES:
Seroprevalence of Varicella-Zoster Virus (VZV) | At Screening Phase (week 0)
Seroprevalence of Herpes Virus-2 (HSV-2) | At Screening Phase (week 0)
Seroprevalence of Cytomegalovirus (CMV) | At Screening Phase (week 0)
Seroprevalence of Epstein Barr (EBV) | At Screening Phase (week 0)
Correlation between the expression of immune activation markers in blood and mucosal tissues | Longidudinally througout the study (up to 12 months)
Correlation between mucosal VZV-specific immune responses and mucosal immune activation | Longidudinally througout the study (up to 12 months)
Acceptability and feasibility of mucosal sampling assessed by participant questionnaires | At study termination - week 50 (+/- 3 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Jaoko, MD, Principal Investigator — KAVI-Institute of Clinical Research / University of Nairobi; Kelly MacDonald, MD, Principal Investigator — University of Toronto; Omu Anzala, MD, Principal Investigator — KAVI-Institute of Clinical Research / University of Nairobi
Locations (1):
- KAVI-ICR, University of Nairobi, Nairobi, Kenya

REFERENCES:
- [Derived] Perciani CT, Farah B, Kaul R, Ostrowski MA, Mahmud SM, Anzala O, Jaoko W; KAVI-ICR Team; MacDonald KS. Live attenuated varicella-zoster virus vaccine does not induce HIV target cell activation. J Clin Invest. 2019 Feb 1;129(2):875-886. doi: 10.1172/JCI124473. Epub 2019 Jan 22. PMID 30511963
- [Derived] Perciani CT, Sekhon M, Hundal S, Farah B, Ostrowski MA, Anzala AO, McKinnon LR, Jaoko W, MacDonald KS; Institute of Tropical and Infectious Diseases (UNITID) Group and the Kenyan AIDS Vaccine Initiative-Institute of Clinical Research (KAVI-ICR) Team. Live Attenuated Zoster Vaccine Boosts Varicella Zoster Virus (VZV)-Specific Humoral Responses Systemically and at the Cervicovaginal Mucosa of Kenyan VZV-Seropositive Women. J Infect Dis. 2018 Sep 8;218(8):1210-1218. doi: 10.1093/infdis/jiy320. PMID 29800309
- [Derived] Perciani CT, Jaoko W, Walmsley S, Farah B, Mahmud SM, Ostrowski M, Anzala O, Team KI, MacDonald KS. Protocol of a randomised controlled trial characterising the immune responses induced by varicella-zoster virus (VZV) vaccination in healthy Kenyan women: setting the stage for a potential VZV-based HIV vaccine. BMJ Open. 2017 Sep 21;7(9):e017391. doi: 10.1136/bmjopen-2017-017391. PMID 28939581